CLINICAL TRIAL: NCT05568095
Title: A Randomized, Open-Label, Multicenter Phase 3 Trial of Domvanalimab, Zimberelimab, and Chemotherapy Versus Nivolumab and Chemotherapy in Participants With Previously Untreated Locally Advanced Unresectable or Metastatic Gastric, Gastroesophageal Junction, and Esophageal Adenocarcinoma
Brief Title: A Clinical Trial of a New Combination Treatment, Domvanalimab and Zimberelimab, Plus Chemotherapy, for People With an Upper Gastrointestinal Tract Cancer That Cannot be Removed With Surgery That Has Spread to Other Parts of the Body
Acronym: STAR-221
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR-221; jRCT2051220179 (Registry Identifier: Japan Registry of Clinical Trials); MOH_2023-04-30_012590 (Registry Identifier: Israel Clinical Research Site - MyTrials); CTR20233469 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform); CTR20233470 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform); 2023-507522-16-00 (Other: EMA: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Advanced Upper Gastrointestinal Tract Adenocarcinoma
Keywords: Domvanalimab; Zimberelimab; Nivolumab; Advanced upper gastrointestinal tract adenocarcinoma; Gastroesophageal junction cancer; Esophageal adenocarcinoma; Gastric cancer; Gastric adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms | interventions — zimberelimab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Domvanalimab + Zimberelimab + FOLFOX/CAPOX (PI Choice) (Experimental): Participants in this arm will receive Domvanalimab and zimberelimab doses once every 4 weeks (Q4W) in addition to chemotherapy with FOLFOX (oxaliplatin, leucovorin, fluorouracil) once every 2 weeks (Q2W) or Domvanalimab and zimberelimab once every 3 weeks (Q3W) in addition to chemotherapy with CAPOX (capecitabine and oxaliplatin) Q3W.
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Capecitabine; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- Nivolumab + FOLFOX/CAPOX (PI Choice) (Active Comparator): Participants in this arm will receive Nivolumab Q2W and FOLFOX Q2W or Nivolumab Q3W + CAPOX Q3W.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Nivolumab

INTERVENTIONS:
Drug: Domvanalimab — Intravenous (IV) Aqueous Solution
  Other Names: AB154
  Arms: Domvanalimab + Zimberelimab + FOLFOX/CAPOX (PI Choice)
Drug: Zimberelimab — IV Aqueous Solution
  Other Names: AB122
  Arms: Domvanalimab + Zimberelimab + FOLFOX/CAPOX (PI Choice)
Drug: Capecitabine — Oral Tablets
Drug: Fluorouracil — IV Aqueous Solution
Drug: Leucovorin — IV Aqueous Solution
Drug: Oxaliplatin — IV Aqueous Solution
Drug: Nivolumab — IV Aqueous Solution
  Arms: Nivolumab + FOLFOX/CAPOX (PI Choice)

SUMMARY:
This randomized Phase 3 open-label study will compare the efficacy of the T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT) monoclonal antibody domvanalimab, the anti programmed cell death protein 1 (PD-1) monoclonal antibody zimberelimab, and multiagent chemotherapy versus the anti PD-1 monoclonal antibody nivolumab and multiagent chemotherapy in the first-line treatment of participants with locally advanced unresectable or metastatic gastric, gastroesophageal junction (GEJ), and esophageal adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of giving signed informed consent which is in compliance with the requirements and restrictions listed in the informed consent form (ICF) and in protocol.
* Histologically confirmed diagnosis of locally advanced unresectable or metastatic gastric, GEJ, or esophageal adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* At least one measurable target lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Key Exclusion Criteria:

* Underlying medical or psychiatric conditions that, in the investigator's or sponsor's opinion, will make the administration of study-specified therapy hazardous, including but not limited to:
* Interstitial lung disease, including history of interstitial lung disease or non-infectious pneumonitis. Active viral, bacterial, or fungal infections requiring parenteral treatment within 14 days of randomization.
* Clinically significant cardiovascular disease, such as New York Heart Association Class II or greater cardiac disease or cerebrovascular accident within 3 months prior to randomization, unstable angina, or new onset angina within 3 months prior to randomization, myocardial infarction within 6 months prior to randomization, or unstable arrhythmia within 3 months prior to randomization.
* History of prior solid-organ transplantation, including allogenic bone marrow transplantation.
* Dementia, psychiatric, or substance abuse disorders that would interfere with satisfying the requirements of the trial.
* Known human epidermal growth factor receptor 2 (HER-2) positive tumor.
* Known untreated, symptomatic, or actively progressing central nervous system (CNS) (brain) metastases. Participants with leptomeningeal metastases are excluded from enrollment.
* Received prior systemic treatment for locally advanced unresectable or metastatic gastric, GEJ, or esophageal adenocarcinoma.
* Disease progression within 6 months of completion of neoadjuvant or adjuvant therapy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until date of death from any cause (Approximately 15 months)]

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization to date of the first documentation of disease progression or date of death from any cause, whichever comes first (Approximately 15 months)
Objective response rate (ORR) | Proportion of randomized participants who achieved a confirmed best overall response of complete response (CR) or partial response (PR) (Approximately 15 months)
Duration of response (DOR) | From the date of first confirmed response (CR or PR), until the date of first documented disease progression or date of death from any cause, whichever comes first (Approximately 15 months)
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From on or after the date of first dose of any study treatment to the date of last study treatment specific safety follow-up or date of initiation of subsequent systemic anti-cancer therapy, whichever occurs first (Approximately 15 months)
Time to first symptom deterioration in the FACT-Ga gastric cancer subscale. | From the date of randomization to change from baseline in subscale greater than or equal to the deterioration threshold, or death from any cause, whichever comes first (Approximately 15 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (205):
- United States (39):
  - Genesis Cancer Center and Blood Institute - Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - UCLA Health - Santa Monica Cancer Care, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - SCRI - Florida Cancer Specialists - South Region Research Office, Fort Myers, Florida
  - SCRI - Florida Cancer Specialists - North Region Research Office, St. Petersburg, Florida
  - SCRI - Florida Cancer Specialists - Panhandle Research Office, Tallahassee, Florida
  - SCRI - Florida Cancer Specialists - East Region Research Office, West Palm Beach, Florida
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute - Poplar Level Road, Louisville, Kentucky
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - HealthPartners Cancer Center at Regions Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Louis Park, Minnesota
  - Perlmutter Cancer Ctr NYU, Mineola, New York
  - Perlmutter Cancer Center - 38th Street, New York, New York
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clin - Fairview Hosp, Cleveland, Ohio
  - Mark H. Zangmeister Cancer Center, Columbus, Ohio
  - Cleveland Clin-Hillcrest Hosp, Mayfield Heights, Ohio
  - Prov Care Clinic - Westside, Portland, Oregon
  - Providence Cancer Center Oncology and Hematology Care Westside Portland, Portland, Oregon
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga - Memorial Plaza, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Centennial, Nashville, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Center for Cancer & Blood Disorders - Fort Worth, Fort Worth, Texas
  - Harris Health System, Houston, Texas
  - USOR - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Fred Hutchinson Cancer Center - Seattle Cancer Care Alliance (SCCA) Location, Seattle, Washington
  - Froedtert Clinical Cancer Center, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Británico de Buenos Aires, Buenos Aires
  - CORI, La Rioja
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
- Australia (4):
  - Monash University, Clayton
  - Gosford Hospital, Gosford
  - Liverpool Hospital, Liverpool
  - Oncology West - Murdoch, Murdoch
- Brazil (5):
  - Fundação Pio XII - Hospital de Câncer de Barretos - Hospital de Amor, Barretos
  - ONCOSITE - Centro de Pesquisa Clinica Em Oncologia Ltda., Ijuí
  - Liga Contra o Câncer - Centro Avançado de Oncologia, Natal
  - Hospital Ernesto Dornelles, Porto Alegre
  - Instituto Nacional de Câncer - Brazil, Rio de Janeiro
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre-Victoria General, Halifax
  - Hôpital Notre-Dame, Montreal
  - Ottawa Hospital - General Campus, Ottawa
  - Princess Margaret Cancer Centre, Toronto
  - Sunnybrook Health Sciences Centre - Bayview Campus, Toronto
- Chile (7):
  - Icegclinic, La Florida
  - Hospital Puerto Montt, Port Montt
  - Oncovida - Santiago, Providencia
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - Centro de Estudios Clínicos SAGA, Santiago
  - Pontificia Universidad Catolica de Chile - Escuela De Medicina - Clinica UC San Carlos de Apoq, Santiago
  - Clínica Universidad Católica del Maule - Talca, Talca
- China (10):
  - Guangdong PR People's Hospital, Guangzhou
  - Sun Yat-Sen Cancer Center, Guangzhou
  - Hainan General Hospital, Haikou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shanghai East Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Qinghai UNV Afl Hospital, Xining
  - Henan Cancer Hospital, Zhengzhou
- France (11):
  - Institut Bergonié, Bordeaux
  - Hôpital Morvan, Brest
  - Centre de Lutte contre le Cancer - François Baclesse, Caen
  - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Armoricain de Radiothérapie, d'Imagerie Médicale et d'Oncologie, Plérin
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Georgia (5):
  - Evex Hospitals - Kutaisi Referral Hospital, Kutaisi
  - LLC Todua Clinic, Tbilisi
  - Ltd Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
  - New Vision University Hospital, Tbilisi
  - Multi-profile Clinic "New Hospitals", Tbilisi
- Guatemala (5):
  - Clínica Privada Dr. Rixci Ramírez, Guatemala City
  - Grupo Medico Angeles, Guatemala City
  - INTEGRA Cancer Institute, Guatemala City
  - Medi-k Cayalá, Guatemala City
  - Centro Regional de Sub Especialidades Médicas (CRESEM) SA, Quetzaltenango
- Hong Kong (4):
  - Hong Kong Sanatorium and Hosp, Happy Valley
  - Humanity & Health Clinical Trial Centre, Hong Kong
  - Queen Mary Hospital - Hong Kong, Hong Kong
  - Tuen Mun Hospital, Tuenmen
- Hungary (4):
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Bács-Kiskun Megyei Oktatókórház - Kecskemét, Kecskemét
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
- Israel (4):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Davidoff Cancer Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Santa Maria Croci, Ravenna
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Rozzano
  - Azienda Sanitaria Universitaria Friuli Centrale ? P.O. Santa Maria della Misericordia, Udine
- Japan (18):
  - Hyogo Cancer Center, Akashi
  - Tokyo Metro Ctr, Bunkyō City
  - University of Tokyo Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Kyushu Cancer Center, Fukuoka
  - Nat Cancer Ctr-Kashiwa Campus, Kashiwa-shi
  - St. Marianna Uni Hosp, Kawasaki
  - Cancer Inst Hosp of JFCR, Kōtō City
  - Kumamoto University Hospital, Kumamoto
  - Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Prefectural Hosp Org, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - Gunma Prefectural Cancer Ctr, Ota-shi
  - Saitama Cancer Center, Saitama
  - National Cancer Ctr Hosp, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Lithuania (4):
  - Kauno Klinikos, Kaunas
  - Klaipedos Universitetine Ligonine, Klaipėda
  - Nacionalinis Vėžio Institutas, Vilnius
  - Vilniaus Universiteto Ligoninė Santariškių Klinikos, Vilnius
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pusat Perubatan Universiti Malaya, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
- Mexico (5):
  - CLIMERS Clinical Medical Research, Colonia Centro
  - Centro Especializado en Investigacion y Tratamiento Oncologicos SC, Mexico City
  - Centro de Atención e Investigación Clínica en Oncología, Mérida
  - Hospital Zambrano Hellion TecSalud, San Pedro Garza García
  - Centro Hemato - Oncológico Privado (CHOP), Toluca
- Peru (4):
  - Hosp Nacional Daniel Carrion, Bellavista
  - SANNA - Clínica El Golf, San Isidro
  - Hospital Maria Auxiliadora, San Juán de Miraflores
  - Instituto Nacional de Enfermedades Neoplásicas, Surquillo
- Philippines (4):
  - Dr Pablo O. Torre Memorial Hospital - Riverside Medical Center, Bacolod City
  - Baguio General Hospital and Medical Center, Baguio City
  - Cebu Doctors' University Hospital, Cebu City
  - Manila Doctors Hospital, Manila
- Poland (4):
  - Centrum Onkologii Ziemi Lubelskiej im. św. Jana z Dukli, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Szpital Miejski w Tychach, Tychy
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Fundação D. Anna de Sommer Champalimaud e Dr. Carlos Montez Champalimaud, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, Porto
- Romania (8):
  - Spitalul Judetean de Urgenta, Baia Mare
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - Medisprof, Cluj-Napoca
  - Centrul De Oncologie Sf Nectarie, Craiova
  - Centrul de Radioterapie Amethyst Cluj, Florești
  - Centrul de Oncologie Euroclinic, Iași
  - Clinica SIGMedical, Suceava
- Serbia (3):
  - Institute of Oncology and Radiology of Serbia (Institut za onkologiju i radiologiju Srbije), Belgrade
  - University Hospital Medical Center (KBC) Bezanijska Kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- South Korea (8):
  - Dong-A University Hospital, Busan
  - Kyungpook Nat Uni Chilgok, Daegu
  - Cha Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Nat Uni Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (8):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital, Bang Phlat
  - Songklanagarind Hospital, Hat Yai
  - Sunpasitthiprasong Hospital, Ubon Ratchathani
- Turkey (Türkiye) (10):
  - T.C. Saglik Bakanligi Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Trakya Universitesi Tip Fakultesi, Edirne
  - T.C. Saglik Bakanligi - Istanbul Il Saglik Mudurlugu - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Kocaeli Üniversitesi Araştırma ve Uygulama Hastanesi, İzmit
  - Inönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
  - Ankara Üniversitesi Tıp Fakültesi - Cebeci Araştırma ve Uygulama Hastanesi, Mamak
  - Van Yüzüncü Yıl Üniversitesi Dursun Odabaş Tıp Merkezi, Van
  - Ataturk Universitesi Arastirma Hastanesi, Yakutiye
  - Başkent Üniversitesi Adana Dr Turgut Noyan Uygulama ve Araştirma Merkezi, Yüreğir
- United Kingdom (7):
  - Barts Health NHS Trust, London
  - Sarah Cannon Research Institute London, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents [e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)] upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: STAR-221 Public Website — https://trials.arcusbio.com/study/?id=STAR-221